CLINICAL TRIAL: NCT02764320
Title: Determining the Optimal Treatment Strategy for Patients Who Have Chronic Migraine With Medication Overuse
Brief Title: The MOTS (Medication Overuse Treatment Strategy) Trial
Acronym: MOTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Todd J. Schwedt, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-001036; PCORI (Other Grant/Funding Number: PCS-1504-30133)
Record Dates: First submitted 2016-05-04; First posted 2016-05-06 (Estimated); Results first posted 2021-11-12 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Discontinuation (Active Comparator): Migraine prophylactic therapy will be initiated or optimized with the immediate discontinuation of the overused medication(s)
  Interventions: Other: Discontinuation of Overused Medication
- Preventive Therapy Only (Active Comparator): Migraine prophylactic therapy will be initiated or optimized without the early discontinuation of the overused medication(s)
  Interventions: Other: Migraine Prophylactic Therapy Only

INTERVENTIONS:
Other: Migraine Prophylactic Therapy Only — Start of new migraine preventive therapy or adjustment of current preventive therapy without immediate discontinuation of the overused medication(s)
  Arms: Preventive Therapy Only
Other: Discontinuation of Overused Medication — Immediate discontinuation of the overused medication(s) and the start of new migraine preventive therapy or adjustment of current preventive therapy
  Arms: Discontinuation

SUMMARY:
There are two commonly used treatment strategies for treating patients who have chronic migraine with medication overuse. This study will compare the outcomes amongst patients randomized to one of the two treatment strategies.

ELIGIBILITY:
Inclusion Criteria

* Adults, at least 21 years of age
* Chronic Migraine - diagnosed according to ICHD3beta criteria
* Medication Overuse - diagnosed according to ICHD3beta criteria
* Willingness to be randomized to either of the two treatment arms
* Willingness to maintain a headache diary
* Plan for follow-up care with the clinician
* No changes to migraine prophylactic therapy within the 4 weeks prior to randomization.

Exclusion Criteria

* Younger than 21 years of age
* Headache diagnoses other than chronic migraine with medication overuse; episodic tension-type headache on 3 or fewer days per month is allowed
* Not willing to be randomized to either of the treatment arms
* Not willing to maintain a daily headache diary
* Not planning on follow-up care with the clinician
* In the opinion of the clinician, randomization to either treatment arm would be considered unsafe (ex: pregnancy, immediate discontinuation
* Prisoners
* Diminished decision-making capacity which in the investigator's opinion would interfere with the person's ability to provide informed consent and complete study procedures.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd J Schwedt, MD, Principal Investigator — Mayo Clinic; David W Dodick, MD, Principal Investigator — Mayo Clinic
Locations (29):
- United States (29):
  - Northern Arizona Healthcare Medical Group, Flagstaff, Arizona
  - Mayo Clinic in Arizona Headache Center, Phoenix, Arizona
  - Mayo Clinic in Arizona Neurology Center, Phoenix, Arizona
  - Honor Health Neurology, Scottsdale, Arizona
  - Mayo Clinic Thunderbird, Scottsdale, Arizona
  - Keck Medical Center of USC, Los Angeles, California
  - University of Colorado Denver Headache Center, Aurora, Colorado
  - University of Colorado Denver Primary Center, Denver, Colorado
  - Blue Sky Neurology, Greenwood Village, Colorado
  - Memorial Healthcare, Hollywood, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Norton Neurology, Louisville, Kentucky
  - Brigham Women's Hospital Headache Clinic, Boston, Massachusetts
  - Brigham Women's Hospital Neurology Clinic, Boston, Massachusetts
  - Henry Ford Allegiance Health, Jackson, Michigan
  - Mayo Clinic Headache Center, Rochester, Minnesota
  - The Headache Center, Ridgeland, Mississippi
  - Clinvest Research, Springfield, Missouri
  - University of Cincinnati Neurology, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Cincinnati Headache Center, Dayton, Ohio
  - Toledo Clinic Adult Neurology, Toledo, Ohio
  - Thomas Jefferson University Hospital Headache Center, Philadelphia, Pennsylvania
  - Preferred Headache Center, Pittsburgh, Pennsylvania
  - University of Utah Primary Care, Salt Lake City, Utah
  - University of Utah General Neurology, Salt Lake City, Utah
  - University of Utah Headache Center, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
  - West Virginia University Neurology, Morgantown, West Virginia

REFERENCES:
- [Derived] Whitaker DJ, Dumkrieger GM, Hentz JG, Dodick DW, Schwedt TJ. Physical impairment during and between migraine attacks: A daily diary study of patients with chronic migraine. Cephalalgia. 2024 Apr;44(4):3331024241249747. doi: 10.1177/03331024241249747. PMID 38663902
- [Derived] Schwedt TJ, Hentz JG, Sahai-Srivastava S, Murinova N, Spare NM, Treppendahl C, Martin VT, Birlea M, Digre K, Watson D, Leonard M, Robert T, Dodick DW; MOTS Investigators. Patient-Centered Treatment of Chronic Migraine With Medication Overuse: A Prospective, Randomized, Pragmatic Clinical Trial. Neurology. 2022 Apr 5;98(14):e1409-e1421. doi: 10.1212/WNL.0000000000200117. Epub 2022 Feb 15. PMID 35169011
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Discontinuation | Preventive Therapy Only
Started | 361 | 359
Completed | 310 | 310
Not Completed | 51 | 49
Not completed — Withdrawal by Subject | 35 | 38
Not completed — Protocol Violation | 11 | 6
Not completed — Adverse Event | 2 | 0
Not completed — Health Issues unable to continue | 2 | 0
Not completed — Did not meet inclusion criteria | 1 | 0
Not completed — Subject moved | 0 | 2
Not completed — Overused medication unavailable | 0 | 1
Not completed — Seeking care outside site | 0 | 1
Not completed — Technology barriers | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Discontinuation | Preventive Therapy Only | Total
Number analyzed (Participants) | 361 | 359 | 720
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (13) | 44 (13) | 44 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 313 | 317 | 630
  Male | 48 | 42 | 90
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 270 | 273 | 543
  Other | 91 | 86 | 177
Region of Enrollment [Number; unit: participants]
  United States | 361 | 359 | 720

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Moderate to Severe Headache Days
Description: Number of days on which a headache lasts for at least 2 hours and at any time peaks at moderate or severe intensity
Time Frame: 12 weeks
Population: Data not collected or analyzed on 16 subjects from the discontinuation arm. Data not collected or analyzed on 19 subjects from the preventive therapy only arm.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Discontinuation | Preventive Therapy Only
Number analyzed (Participants) | 294 | 291
days | 9.3 (7.2) | 9.1 (6.8)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study for a total of approximately 48 weeks on all participants.
Arm/Group | Discontinuation | Preventive Therapy Only
All-Cause Mortality (participants affected / at risk) | 0/361 | 1/359
Serious Adverse Events (participants affected / at risk) | 7/361 | 7/359
Other Adverse Events (participants affected / at risk) | 20/361 | 16/359
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Discontinuation (N=361) | Preventive Therapy Only (N=359)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Cecal Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Headache Worsened (Nervous system disorders) | 1 (1) | 0 (0)
Joint Range of Motion Decrease Cervical Spine (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Surgical Procedure - Spine (Surgical and medical procedures) | 1 (1) | 0 (0)
Thromboembolic Event (Vascular disorders) | 0 (0) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Discontinuation (N=361) | Preventive Therapy Only (N=359)
Fatigue (General disorders) | 4 (4) | 2 (2)
Sinusitis (Infections and infestations) | 4 (4) | 0 (0)
Weight Gain (Investigations) | 1 (1) | 6 (6)
Headache Worsened (Nervous system disorders) | 6 (6) | 5 (5)
Paresthesia (Nervous system disorders) | 7 (7) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT02764320/Prot_SAP_000.pdf